CLINICAL TRIAL: NCT05661370
Title: Improving Diagnostic Accuracy in Skin Cancer Diagnostics Using Educational Mobile App: a Randomized Controlled Study
Brief Title: App Teaches Doctors to Diagnose Skin Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Gustav Gede Nervil, Medical Doctor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GP-Learn
Record Dates: First submitted 2022-12-05; First posted 2022-12-22 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Melanoma (Skin); Carcinoma
Keywords: Digital Learning; e-learning; Melanoma; Carcinoma; Dermoscopy; Dermloop
MeSH Terms: conditions — Melanoma; Carcinoma

STUDY DESIGN:
Intervention Model Description: Intervention and Controlgroup parallel design using sequential continues block randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Access to educational mobile application for 8 days, diagnosing 500 digital patient-cases.
  Interventions: Other: Dermloop Learn
- Control (No Intervention): Control group receiving no intervention, continuing daily practice.

INTERVENTIONS:
Other: Dermloop Learn — Educational Mobile Application with a library of digital patient-cases and written learning modules the user can access on 36 common skin lesions, both benign and malignant.
  Arms: Intervention

SUMMARY:
This study aimed to examine if self-paced learning with a novel digital patient-case-based educational platform can increase primary care physicians' diagnostic accuracy of malignant and benign skin lesions on both the level of benign/malignant and the diagnosis level. Secondarily the study aimed to investigate the time spent in reaching this change in proficiency.

DETAILED DESCRIPTION:
Participants were given a questionnaire and an initial Skin Cancer Multiple Choice-Questionnaire (MCQ) to test their diagnostic skills regardining skin and mole cancer and the most common differential diagnoses.

Participants in the Intervention group was then given access to an educational mobile application (App) for 8 days and asked to diagnose 500 patient cases. The participants did so at their own leisure and time.

After 8 days they were asked to abstain from using the App for another 8 days (wash out period) and were then given a Final Skin Cancer Multiple Choice-Questionnaire (MCQ).

Participants of the control group received no intervention nor education during the 16 days of waiting before they took the final Skin Cancer Multiple Choice-Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Physician who works in General Practice

Exclusion Criteria:

-

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Multiple-Choice Questionnaire (MCQ) Score | Before and immediately after intervention (On average 19 days after enrollment)
  Participants are given a test before and after the intervention using a skin cancer MCQ test with 12 digital-patient cases. A higher score means better diagnostic proficiency. The primary outcome is the change of this score.

SECONDARY OUTCOMES:
Diagnostic proficiencies | During the 8 days of access to the educational mobile application.
  Sensitivity, Specificity and Positive Predictive Value of the participants in the intervention group, calculated on their cases seen in the educational mobile application.
Time spend | During the 8 days of access to the educational mobile application.
  The Dermloop Learn app tracks how much time each user spends quizzing and reading.

CONTACTS AND LOCATIONS:
Locations (1):
- AISC Research Fascility, Copenhagen, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Participant quiz-answer data can be shared upon reasonable request.
Time Frame: After publication
Access Criteria: Researchers with interest in skin cancer diagnostics.
URL: https://aiscresearch.com/

REFERENCES:
- [Derived] Nervil GG, Ternov NK, Vestergaard T, Solvsten H, Chakera AH, Tolsgaard MG, Holmich LR. Improving Skin Cancer Diagnostics Through a Mobile App With a Large Interactive Image Repository: Randomized Controlled Trial. JMIR Dermatol. 2023 Aug 9;6:e48357. doi: 10.2196/48357. PMID 37624707